CLINICAL TRIAL: NCT02929264
Title: An fMRI Study in Healthy Volunteers to Investigate the Effects of ABX-1431 on Experimental Hyperalgesia and Its Neural Correlates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abide Therapeutics (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ABX-1431_PN003
Record Dates: First submitted 2016-10-03; First posted 2016-10-11 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Pain
Keywords: Healthy volunteer; Experimental hyperalgesia; fMRI
MeSH Terms: conditions — Pain | interventions — ABX-1431

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABX-1431 (Experimental): ABX-1431, capsules, 40 mg, single dose
  Interventions: Drug: ABX-1431
- Placebo (Placebo Comparator): Placebo, capsules, single dose
  Interventions: Drug: Placebo
- Control (No Intervention): No Intervention

INTERVENTIONS:
Drug: ABX-1431 — Capsules, 40 mg, single dose
  Arms: ABX-1431
Drug: Placebo — Capsules, single dose
  Arms: Placebo

SUMMARY:
An fMRI study in healthy volunteers to investigate the effects of ABX-1431 on experimental hyperalgesia and its neural correlates.

ELIGIBILITY:
Inclusion Criteria:

* Understands the study procedures and is willing and able to give informed consent for participation in the trial.
* Male, right-handed, aged 18 to 55 years of age at the first visit.
* Body mass index >18 and ≤30 kg/m2 at the first visit.
* Judged to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests (see appendix A for interpretation of laboratory findings) obtained at the first visit.
* No clinically significant abnormality of ECG performed on the first visit.
* Is a non-smoker and has not used nicotine or nicotine-containing products for at least 3 months.
* In the Investigator's opinion, participant is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner to be notified of participation in the trial and to confirm the eligibility of the participant.
* Able to tolerate MRI scanning at the first visit. Responds to topical capsaicin by attaining a pain score of at least 4/10, assessed on the first visit.

Exclusion Criteria:

* A current acute pain condition.
* A personal history of a chronic pain condition.
* Contraindications to MRI scanning.
* Scheduled elective surgery or other procedures requiring general anesthesia during the trial.
* A personal history of a clinically significant psychiatric disorder (including severe affective disorder, anxiety disorders, psychotic tendencies and drug-induced psychoses). Subjects who have had situational depression in the past may be enrolled at the discretion of the investigator.
* A first-degree family history of schizophrenia, major affective disorder, or other psychosis.
* Participant is mentally or legally incapacitated, has significant emotional problems at the time of the first visit, or is expected to have potential for mental incapacitation during the conduct of the study.
* A history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the participant by virtue of their participation in the study.
* An estimated creatinine clearance of ≤80ml/min based on the Cockcroft-Gault equation. An actual creatinine clearance, as measured using a 24-hour urine collection, may be used in place of, or in conjunction with the Cockcraft-Gault calculation. Subjects with an actual or calculated creatinine clearance that is in the range of 72-79 mL/min (i.e., within 10% of 80 mL/min) may be enrolled in the study at the discretion of the Investigator.
* A history of stroke, chronic seizures, or major neurological disorder.
* A history of clinically significant (in the opinion of the investigator) endocrine, gastrointestinal, cardiovascular, peripheral vascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Participants with history of uncomplicated kidney stones (defined as spontaneous passage and no recurrence in the last 5 years) or childhood asthma may be enrolled in the trial at the discretion of the investigator.
* A history of clinically significant neoplastic disease, with the exception of adequately treated localized or in situ non-melanoma carcinoma of the skin.
* A history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs (including capsaicin and marijuana or other cannabis-containing drugs) or food.
* Participants who have had major surgery or have donated or lost 1 unit (approximately 500ml) of blood within 4 weeks prior to the first visit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Brain activity in response to noxious stimuli, as assessed by fMRI, following a single dose of ABX-1431, compared to the same outcome following placebo and no treatment interventions. | Approximately 5 weeks

SECONDARY OUTCOMES:
Pain scores, assessed by VAS for ongoing and evoked pain, recorded after sensitization with topical 1% capsaicin. Pain scores following single oral doses of ABX-1431 will be compared to those following placebo and no treatment. | Approximately 5 weeks
Severity of, and Number of Participants With Clinical and Laboratory Adverse Events (AE) following single oral doses of ABX-1431, placebo and no treatment as a Measure of Safety and Tolerability. | Approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tracey, DPhil., FRCA, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom